CLINICAL TRIAL: NCT00939458
Title: A Randomized, Open Label, Single Dose, Crossover, Bioequivalence Study of Lamotrigine 2 x 25 mg IR Tablets of Torrent Pharmaceuticals Pvt., Ltd., India and Lamictal ® (Lamotrigine) 2 x 25 mg Tablets of Glaxo-SmithKline, USA, in Healthy Human Adult Subjects,Under Fed Conditions
Brief Title: Study of Lamotrigine 2 x 25 mg IR Tablets of Torrent Pharmaceuticals Pvt., Ltd., India and Lamictal ® (Lamotrigine) 2 x 25 mg Tablets of Glaxo-SmithKline, USA, in Healthy Human Adult Subjects, Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 1087/06
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine

SUMMARY:
* Objective:

  * To assess the bioequivalence of Lamotrigine 2 x 25 mg IR tablets of Torrent Pharmaceuticals Pvt., Ltd., India and Lamictal ® (Lamotrigine) 2 x 25 mg tablets of Glaxo-SmithKline, USA, in healthy human adult subjects, under fed conditions.
* Study Design:

  * A randomized, open label, two treatment, two period, two sequence, single dose, crossover study, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects of either sex between 18-55 years of age (inclusive), having a body mass index (BMI) between 18 and 27 kg/m2
* Subjects who have no evidence of underlying disease during screening and whose physical examination is performed within 21 days prior to commencement of the study.
* Subjects whose screening laboratory values are within normal limits or values outside normal limits considered by the physician/Principal Investigator to be of no clinical significance.
* Informed consent given in written form according to section 11.3 of the protocol.
* Female Subjects:

  1. of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  2. postmenopausal for at least 1 year.
  3. surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

* Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
* Alcohol dependence, alcohol abuse or drug abuse within past one year.
* Moderate to heavy smoking (> 10 cigarettes/day) or consumption of tobacco products.
* History of difficulty in swallowing tablet.
* Clinically significant illness within 4 weeks before the start of the study
* Asthma, urticaria or other allergic type reactions after taking any medication.
* Positive urine drug screening, HIV, Hepatitis B & C tests.
* Any history of hypersensitivity to Lamotrigine.
* Existence of any surgical or medical condition, which, in the judgment of clinical investigator might interfere with the pharmacokinetics of the drug or likely to compromise the safety of the subject.
* Inability to communicate or co-operate with the investigator due to language problem, attitude, poor mental development/impaired cerebral function.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Labs Pvt. Ltd., Bangalore, Karnataka, India